CLINICAL TRIAL: NCT00003916
Title: Focal Fractionated Conformal Stereotactic Boost Following Conventional Radiotherapy of High Grade Gliomas: A Randomized Phase III Study
Brief Title: Standard Radiation Therapy With or Without Stereotactic Radiation Therapy in Treating Patients With Glioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-22972-26991; EORTC-22972; EORTC-26991; MRC-BR10
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — Radiotherapy; Radiosurgery

INTERVENTIONS:
Radiation: radiation therapy
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells and may be an effective treatment for patients with glioma. Stereotactic radiation therapy may be able to deliver x-rays directly to the tumor and cause less damage to normal tissue. It is not yet known if standard radiation therapy is more effective when followed by stereotactic radiation therapy.

PURPOSE: Randomized phase III trial to compare the effectiveness of standard radiation therapy with or without stereotactic radiation therapy in treating patients who have glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of adjuvant conventional radiotherapy with or without fractionated stereotactic boost radiotherapy on survival in patients with high grade glioma. II. Compare the quality of life of these patients after these therapies.

OUTLINE: This is a randomized study. Patients are stratified according to WHO disease grade (III vs IV), center, and age (under 40 vs 40 and over). Patients are randomized to undergo stereotactic radiotherapy or no further treatment after conventional radiotherapy. Patients undergo conventional radiotherapy once or twice a day for up to 6 weeks. Patients randomized to receive additional treatment receive stereotactically guided conformal boost radiotherapy for 4 days, within 4 weeks after completion of conventional radiotherapy. Quality of life is assessed before radiotherapy, then at follow up visits. Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 605 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven WHO grade III or IV glioma at primary diagnosis that enhance on preoperative imaging Glioblastoma Anaplastic astrocytoma Gliosarcoma Tumor volume no greater than 4.0 cm in maximum diameter on preoperative CT or MRI No prior histology of WHO grade I or II glioma Astrocytoma Oligodendroglioma No brainstem or infratentorial tumor No multifocal glioma Safe to treat tumor stereotactically No close proximity to critical structures, e.g., optic chiasm

PATIENT CHARACTERISTICS: Age: 18 to 65 Performance status: WHO 0 or 1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Able to tolerate full course of conventional radiotherapy No prior or concurrent medical condition that would preclude study therapy No prior malignancies within 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy No concurrent adjuvant chemotherapy Endocrine therapy: Concurrent steroids allowed Radiotherapy: See Disease Characteristics No prior radiotherapy to the head and neck area No prior radiotherapy to the brain No more than 6 weeks since other prior radiotherapy Surgery: See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-04; Primary Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta Baumert, MD, PhD, Study Chair — UniversitaetsSpital Zuerich
Locations (8):
- Alfred Hospital, Melbourne, Victoria, Australia
- Centre Antoine Lacassagne, Nice, France
- Germany (2):
  - Medizinische Klinik I, Dresden
  - Universitaet Wuerzburg/Hautkrankheiten, Würzburg
- Vrije Universiteit Medisch Centrum, Amsterdam, Netherlands
- Institut Catala d'Oncologia - Hospital Duran i Reynals, Barcelona, Spain
- Universitaetsspital, Zurich, Switzerland
- Royal Marsden Hospital, Sutton, England, United Kingdom

REFERENCES:
- [Result] Baumert BG, Brada M, Bernier J, Kortmann RD, Dehing-Oberije C, Collette L, Davis JB. EORTC 22972-26991/MRC BR10 trial: fractionated stereotactic boost following conventional radiotherapy of high grade gliomas. Clinical and quality-assurance results of the stereotactic boost arm. Radiother Oncol. 2008 Aug;88(2):163-72. doi: 10.1016/j.radonc.2008.03.025. Epub 2008 Apr 30. PMID 18455252
- [Result] Brada M, Baumert B. Focal fractionated conformal stereotactic boost following conventional radiotherapy of high-grade gliomas: a randomized phase III study. A joint study of the EORTC (22972) and the MRC (BR10). Front Radiat Ther Oncol. 1999;33:241-3. doi: 10.1159/000061233. No abstract available. PMID 10549493